CLINICAL TRIAL: NCT03710473
Title: Non-invasive and Continuous Monitoring of Diastolic Blood Pressure: a Prospective Observational Study - IMPACT
Brief Title: Non-Invasive Blood Pressure Measurement in Critically Ill PAtients Post Cardiosurgical Therapy
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Ava AG (Industry); CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Other Study IDs: HOPE CT 1
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Systemic Hypertension
Keywords: Hypertension; Non-invasive blood pressure Monitoring; Photoplethysmography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optical sensor, Pulse watch — Continuous blood pressure monitoring obtained by a Pulse watch

SUMMARY:
The aim of the present study is to evaluate the accuracy of measuring beat-by-beat diastolic blood pressure from a non-invasive, cuffless and non-obtrusive watch-like optical device worn at the wrist.

DETAILED DESCRIPTION:
Given the prevalence of hypertension in society and the current limitations associated with oscillometric cuffs, the need for a continuous cuffless alternative for blood pressure home monitoring at a global scale is paramount. Such a device would not only improve the global control of blood pressure, but more generally, it could have a larger social impact by improving the comfort and reducing the stress for the clinical management of hypertensive patients.

In the present study the investigators seek to investigate, as a primary purpose, to evaluate the accuracy of non-invasive blood pressure measurements via a watch-like optical sensor and compare these to standard monitoring (arterial line).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cardiac or vascular surgery, with presence of a radial arterial line for perioperative management;
* Willing and able to provide Informed Consent.

Exclusion Criteria:

* (Chronic) pace-maker/ defibrillator in situ at study inclusion;
* Known severe aortic stenosis (mean gradient > 40 mmHg, valve area < 1 cm2);
* Rhythmogenic heart disease (resting heart rate > 120/min) at time of study inclusion;
* Emergency patient (i.e. unscheduled OR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled for cardiac or vascular surgery at the Department of Cardiovascular Surgery of Inselspital, Bern.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of diastolic blood pressures (in mmHg) assessed via non-invasive vs. invasive blood pressure (arterial line) measurement | 24 hours
  Statistical comparison of both measures of diastolic blood pressure

SECONDARY OUTCOMES:
Descriptive assessment: time until normalization of measurement after re-calibration of diastolic blood pressure measurement using the non-invasive approach | 24 hours
  To evaluate the influence of the re-calibration time interval (amount of time in-between two consecutive calibrations of the optical devices) on the accuracy of diastolic blood pressure assessment.
Descriptive analysis of comparison to measurements at the fingertip (non-invasive vs. fingertip diastolic blood pressure assessment) | 24 hours
  To compare the accuracy when applied to photoplethysmographic signals measured at the wrist versus signals measured at the fingertip.

CONTACTS AND LOCATIONS:
Overall Officials: David Reineke, MD, Principal Investigator — Dept of Cardiovascular Surgery
Locations (1):
- Inselspital, Dept of Intensive Care Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No